CLINICAL TRIAL: NCT01212029
Title: Testing and Calibration of Non-Invasive Optical Imaging Technology for Functional Brain Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); National Institutes of Health Clinical Center (CC) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 100198; 10-CH-0198
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-10-02

CONDITIONS: Cognition
Keywords: fNIRS; Healthy Volunteer; HV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 1/All Subjects (Experimental): Imaging studies related to functional brain activation
  Interventions: Behavioral: Behavioral measures; Device: fNIRS Devices & Application; Other: Physiological measures

INTERVENTIONS:
Behavioral: Behavioral measures — Behavioral tasks/ questionnaires
Device: fNIRS Devices & Application — Device 1- fNIRSoft and Device 2 - NIRScout
Other: Physiological measures — A set of tasks.

SUMMARY:
Background:

- Non-invasive functional near infrared (fNIR) imaging techniques use infrared light to detect changes in blood volume and oxygen levels during brain activity. fNIR is being studied as a possible way to examine the brain activity of individuals who are unable to undergo standard brain function imaging techniques (such as functional magnetic resonance imaging, or fMRI). For instance, war veterans who have iron shrapnel in the body are not able to have fMRI scans, and very young children or children with autism and related disorders are often not able or willing to cooperate long enough in the MRI environment to allow full imaging studies to take place. Researchers are interested in comparing the results of fNIR and fMRI performed on healthy volunteers to determine if fNIR produces similarly accurate results.

Objectives:

- To examine the capabilities of non-invasive functional near infrared imaging techniques on healthy volunteers and compare the results with the existing outcomes of functional magnetic resonance imaging.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Participants will have one study visit. Depending on the complexity of the task, the whole exam will take between 5 minutes and 1 hour to perform.
* Participants will be asked to sit as still as possible while wearing a headband that includes light sources and detectors (the fNIR device).
* Participants will be asked to perform a set of tasks (e.g., reading sentences or counting numbers in one s head). Data will be collected during these experiments.

DETAILED DESCRIPTION:
Objective: to a) cross-validate our near infrared spectroscopy (NIRS) imaging system with existing functional magnetic resonance imaging (fMRI) and electroencephalogram (EEG) data, and b) to investigate any significant technical issues associated with optode placement and motion artifacts, and to explore techniques that will potentially improve the feasibility and reliability of the system according to the needs of the population for whom existing imaging systems are unsuitable.

Study population: 250 healthy volunteers

Design: The study will look for correlations between NIRS signal changes in healthy subjects when performing functional tasks, and existing fMRI data.

Outcome Measures: graded changes in blood flow and oxygen, measured with NIRS, in response to different functional tasks.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 years or greater.

EXCLUSION CRITERIA:

* Healthy volunteers with any skin disease that, in the opinion of the investigator, would interfere with the study measurements.
* Healthy volunteers with any past or present vascular disease.
* Known adverse reaction to latex.
* Any medical condition that, in the opinion of the Principal Investigator would preclude the inclusion of a patient onto this research study.
* Unable or unwilling to give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-09-08 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Gandjbakhche, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bozkurt A, Onaral B. Safety assessment of near infrared light emitting diodes for diffuse optical measurements. Biomed Eng Online. 2004 Mar 22;3(1):9. doi: 10.1186/1475-925X-3-9. PMID 15035670
- [Background] Friedland RP, Iadecola C. Roy and Sherrington (1890): a centennial reexamination of "On the regulation of the blood-supply of the brain". Neurology. 1991 Jan;41(1):10-4. doi: 10.1212/wnl.41.1.10. No abstract available. PMID 1985272
- [Background] Villringer A, Chance B. Non-invasive optical spectroscopy and imaging of human brain function. Trends Neurosci. 1997 Oct;20(10):435-42. doi: 10.1016/s0166-2236(97)01132-6. PMID 9347608
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CH-0198.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/All Subjects
Started | 159
Completed | 159
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 6 participants did not report their gender.
Groups:
- All Subjects: Imaging studies related to functional brain activation
Arm/Group | All Subjects
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: year] | 36 (13)
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 30
  White | 77
  More than one race | 3
  Unknown or Not Reported | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 128
  Unknown or Not Reported | 16
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 participants did not report their gender.
  Participants
    number analyzed (Participants) | 153
    Female | 87
    Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Prefrontal Cortex Activation and Respiratory Sinus Arrhythmia
Description: Prefrontal cortex (PFC) activation is measured in term of change in oxyhemoglobin (O2Hb) using a functional Near-Infrared Spectroscopy (fNIRS) system at a person forehead.
  Respiratory Sinus Arrhythmia (RSA) is the variation of heart beat in response to breathing. It is calculated as changes in the lengths of interbeat interval as a result of breathing using root mean square successive difference (RMSSD).
  The relationship between activation of PFC and RSA is quantified as a linear regression coefficient, which represents the estimated average change in O2Hb concentration associated with a 1 unit increase in RMSSD in heartrate interbeat interval length.
Time Frame: During the assessment
Population: Healthy adults (mean age = 37.18 years, SD = 14.67).
Measure: Mean (Standard Deviation); unit: Micro mol per second
Groups:
- Baseline: Relationship between PFC activation and RSA was evaluated during baseline condition, where participants were instructed to sit quietly while watching a mildly stimulating video presented on a computer monitor.
  Data reported is the mean and standard deviation of the regression coefficients of RMSSD predicting O2Hb during baseline across all 16 fNIRS channels at the prefrontal cortex.
- Go/No-Go Task: Relationship between PFC activation and RSA was evaluated during a Go/No-Go task. During the task, participants were instructed to press the space bar in a keyboard when they saw the letter "Y" and not to press any buttons when they saw the letter "X" displayed in a monitor.
  Data reported is the mean and standard deviation of the regression coefficients of RMSSD predicting O2Hb during Go/No-Go task across all 16 fNIRS channels at the prefrontal cortex.
Arm/Group | Baseline | Go/No-Go Task
Number analyzed (Participants) | 38 | 38
Micro mol per second | -0.064 (0.035) | 0.00375 (0.023)
Statistical Analysis 1: Comparison: Baseline; Null hypothesis: there is no significant correlation between RMSSD and O2Hb levels during baseline; Test type: Other — One sample t-tests of standardized regression coefficients of RMSSD predicting O2Hb during baseline; p = 0.008, t-test, 2 sided — t-test was performed 16 times for 16 fNIRS channels. The reported p-value is an uncorrected value for channel 10

2. Primary Outcome: Mean Change in Oxyhemoblobin Concentration in Left Dorsolateral Prefrontal Cortex Region After Impersonal Moral Judgement Dilemma
Description: Moral judgment (MJ) is the process of evaluating what is right or wrong based on social norms. The classic Trolley Dilemma describes an impersonal MJ scenario in which a trolley is hurtling toward five workers on the track. One option presented is to flip a switch to divert the course of the trolley, which would result in the trolley hurtling toward one person on the opposite side of the track, killing this one person. The other is to do nothing and allow the five workers to die.
  Dorsolateral prefrontal cortex (DL-PFC) is responsible for utilitarian (logical) judgments that are thought to engage more cognitive processes and fewer emotional processes.
  Oxyhemoglobin (O2Hb) is measured using a functional Near-Infrared Spectroscopy (fNIRS) at prefrontal cortex.
Time Frame: During the assessment
Population: Healthy participants (15 male, 18 female), aged 18-58 years, with a mean age of 33.7 years.
Measure: Mean (Standard Deviation); unit: Micro mol
Groups:
- Prefrontal Cortex Activation in a Moral Judgment Task Using Functional Near-Infrared Spectroscopy: The study aimed to investigate the neural processes involved in moral judgment (MJ) using fNIRS, focusing on prefrontal cortex activation during emotionally salient (personal) and less emotional (impersonal) moral dilemmas.
Arm/Group | Prefrontal Cortex Activation in a Moral Judgment Task Using Functional Near-Infrared Spectroscopy
Number analyzed (Participants) | 33
Micro mol | 0.0784 (0.0102)
Statistical Analysis 1: Comparison: Prefrontal Cortex Activation in a Moral Judgment Task Using Functional Near-Infrared Spectroscopy; Test type: Other; p = 0.0105, Tukey method

3. Secondary Outcome: Number of Participants With Significant Issues Associated With NIRS
Description: Assess any significant issues associated with NIRS optode placement and evaluate the effect of subject motion on data collection, quality, and noise.
  Data from participants with significant issues, which either due to NIRS optode placement or subject motion, data quality, and noise, are removed from further analysis.
Time Frame: During the assessment
Population: Healthy adults
Measure: Number; unit: participants
Groups:
- Baseline and Go/No-Go Task: Assessment was performed while participants were in a baseline or a Go/No-Go task.
Arm/Group | Baseline and Go/No-Go Task
Number analyzed (Participants) | 44
participants | 6

4. Secondary Outcome: Number of Participants With High Performance But Low Prefrontal Cortex Activation
Description: High performance group include people with accuracy score greater than 90% during an n-back task.
Time Frame: During the assessment
Population: Healthy adults (15 female, 14 male) aged 20-59 years (mean age = 36.2, SD= 12.35).
Measure: Count of Participants; unit: Participants
Groups:
- High Performance Group: Low activation in dorsal lateral prefrontal cortex.
Arm/Group | High Performance Group
Number analyzed (Participants) | 29
Participants | 18

ADVERSE EVENTS:
Time Frame: 1 hour
Groups:
- Neural Effects of Acute Physical Activity on Posture and Inhibitory Control Dual Task: This study investigates neural mechanisms underlying posture-inhibitory control dual-tasking and the acute effects of physical activity on dual-task performance.
Arm/Group | Neural Effects of Acute Physical Activity on Posture and Inhibitory Control Dual Task
All-Cause Mortality (participants affected / at risk) | 0/159
Serious Adverse Events (participants affected / at risk) | 0/159
Other Adverse Events (participants affected / at risk) | 3/159
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neural Effects of Acute Physical Activity on Posture and Inhibitory Control Dual Task (N=159)
Hypertension using CTCAE (General disorders) | 3 (3) — Increase of blood pressure in 3 participants after a 1 minute sit and stand task where a participant alternatively sit and stand continuously for 1 minute.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT01212029/Prot_SAP_000.pdf